CLINICAL TRIAL: NCT04628793
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED, FIRST-IN-HUMAN STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF SINGLE ASCENDING ORAL DOSES OF PF-07258669 ADMINISTERED TO HEALTHY ADULT PARTICIPANTS
Brief Title: A Study of Single Ascending Doses of PF-07258669 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: C4541001; 2020-004280-42 (EudraCT Number)
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Results first posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2023-07

CONDITIONS: Healthy Participants
Keywords: PF-07258669; first in human; melanocortin-4 receptor; MC4R; healthy participants; safety; tolerability; pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Single dose administration of PF-07258669 and placebo; Within a cohort, participants will receive 3 doses of PF-07258669 and 1 dose of placebo.
  Interventions: Drug: PF-07258669; Drug: Placebo
- Cohort 2 (Experimental): Single dose administration of PF-07258669 and placebo; Within a cohort, participants will receive 3 doses of PF-07258669 and 1 dose of placebo.
  Interventions: Drug: PF-07258669; Drug: Placebo
- Cohort 3 (Experimental): Single dose administration of PF-07258669 and placebo; Within a cohort, participants will receive 3 doses of PF-07258669 and 1 dose of placebo.
  Interventions: Drug: PF-07258669; Drug: Placebo

INTERVENTIONS:
Drug: PF-07258669 — PF-07258669 will be prepared as an oral solution and/or suspension given in escalating single doses to be determined
Drug: Placebo — Matching placebo will be prepared as an oral solution and/or suspension given in each cohort

SUMMARY:
This study will be the first time PF-07258669 is administered to humans. The purpose of the study is to evaluate the safety, tolerability, and pharmacokinetics of PF-07258669 following administration of single oral doses to healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Female participants of non-child bearing potential and male participants and who are overtly healthy as determined by medical evaluation including medical history, physical examination, neurological examination, laboratory tests, and cardiac monitoring.
* Participants who are willing to avoid direct sunlight exposure or any high intensity ultraviolet light exposure from admission to the follow-up contact and to apply sunscreen/lotion with a high sun protection factor, as appropriate.
* BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing), as well as presence of lipid panel abnormalities (eg, hypercholesterolemia, hypertriglyceridemia).
* Evidence of history of orthostatic hypotension or symptomatic bradycardia.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
* Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
* Current findings or documented past history of blood pressure values <90 mmHg systolic or <50 mmHg diastolic.
* Any lipid panel parameter (ie, total cholesterol, triglycerides, HDL, and/or LDL) ≥1.25× ULN.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- QPS-MRA, LLC-Main Office, South Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4541001

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Participants in Cohort 1 underwent 4 treatment periods receiving up to 3 doses of PF-07258669 and up to 1 dose of placebo at 0.1mg, 0.3mg, 1mg, and 3mg on Day 1 in Periods 1-4 respectively. There was a washout interval of at least 7 days after each period. At each dose level, participants were assigned in an approximately 3:1 manner to receive PF-07258669 and placebo.
- Cohort 2: Participants in Cohort 2 underwent 4 treatment periods receiving up to 3 doses of PF-07258669 and up to 1 dose of placebo on Day 1 at 10mg, 30mg, 100mg, and 200mg in Periods 1-4 respectively. There was a washout interval of at least 7 days after each period. At each dose level, participants were assigned in an approximately 3:1 manner to receive PF-07258669 and placebo.
- Cohort 3: Participants in Cohort 3 underwent 1 treatment period and received 300 mg PF-07258669 or placebo in a 3:1 manner on Day 1 in Period 1.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 10 (8 participants were planned for all periods in Cohort 1. However, additional participants were enrolled if <8 participants were enrolled in Period 1 and/or to replace participants who dropped out during the study for reasons not related to safety or tolerability. These additional participants may have entered later periods directly.) | 11 (8 participants were planned for all periods in Cohort 2. However, additional participants were enrolled if <8 participants were enrolled in Period 1 and/or to replace participants who dropped out during the study for reasons not related to safety or tolerability. These additional participants may have entered later periods directly.) | 8
Period 1 | 7 (2 participants received placebo and 5 received PF-07258669 0.1mg on Period 1 Day 1.) | 8 (2 participants received placebo and 6 received PF-07258669 10mg on Period 1 Day 1.) | 8 (2 participants received placebo and 6 received PF-07258669 300mg on Period 1 Day 1.)
Period 2 | 7 (2 participants received placebo and 5 received PF-07258669 0.3mg on Period 2 Day 1.) | 7 (2 participants received placebo and 5 received PF-07258669 30mg on Period 2 Day 1.) | 0 (No participant entered Period 2.)
Period 3 | 8 (2 participants received placebo and 6 received PF-07258669 1mg on Period 3 Day 1.) | 8 (2 participants received placebo and 6 received PF-07258669 100mg on Period 3 Day 1.) | 0 (No participant entered Period 3.)
Period 4 | 8 (2 participants received placebo and 6 received PF-07258669 3mg on Period 4 Day 1.) | 8 (2 participant received placebo and 6 received PF-07258669 200mg on Period 4 Day 1.) | 0 (No participant entered Period 4.)
Completed (Completion of the entire study including the follow-up phase) | 8 | 7 (1 participant completed double blind treatment and discontinued during follow-up phase due to lost to follow-up.) | 0
Not Completed | 2 | 4 | 8
Not completed — Study terminated by sponsor | 0 | 0 | 8
Not completed — Withdrawal by Subject | 2 | 3 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received a dose of study intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 10 | 11 | 8 | 29
Age, Continuous [Median (Full Range); unit: Years] | 39.5 [23.0 to 54.0] | 42.0 [34.0 to 52.0] | 32.5 [20.0 to 56.0] | 40.0 [20.0 to 56.0]
Age, Customized [Count of Participants; unit: Participants]
  18-44 Years | 6 | 8 | 5 | 19
  45-60 Years | 4 | 3 | 3 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 4 | 9
  Male | 7 | 9 | 4 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 10 | 7 | 26
  Black or African American | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical study subject, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A serious AE (SAE) was defined as any untoward medical occurrence that, at any dose: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent disability/incapacity; was a congenital anomaly/birth defect; or other serious situations such as important medical events. TEAEs were events between first dose of study drug and up to follow-up visit that were absent before treatment or that worsened after treatment. AEs presented below were TEAEs. The investigator was required to use clinical judgment to assess the potential relationship between investigational product and each AE, to define an treatment-related AE.
Time Frame: From first dose of study intervention (Day 1) to telephone Follow Up (28-35 days after lase dose of study intervention) (approximately up to 20 weeks)
Population: The safety analysis set included all participants randomly assigned to study intervention and who received a dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Placebo: All participants who received placebo in any period of any cohort
- PF-07258669 0.1mg: Participants in Cohort 1 who received PF-07258669 0.1mg
- PF-07258669 0.3mg: Participants in Cohort 1 who received PF-07258669 0.3mg
- PF-07258669 1mg: Participants in Cohort 1 who received PF-07258669 1mg
- PF-07258669 3mg: Participants in Cohort 1 who received PF-07258669 3mg
- PF-07258669 10mg: Participants in Cohort 2 who received PF-07258669 10mg
- PF-07258669 30mg: Participants in Cohort 2 who received PF-07258669 30mg
- PF-07258669 100mg: Participants in Cohort 2 who received PF-07258669 100mg
- PF-07258669 200mg: Participants in Cohort 2 who received PF-07258669 200mg
- PF-07258669 300mg: Participants in Cohort 3 who received PF-07258669 300mg
Arm/Group | Pooled Placebo | PF-07258669 0.1mg | PF-07258669 0.3mg | PF-07258669 1mg | PF-07258669 3mg | PF-07258669 10mg | PF-07258669 30mg | PF-07258669 100mg | PF-07258669 200mg | PF-07258669 300mg
Number analyzed (Participants) | 18 | 5 | 5 | 6 | 6 | 6 | 5 | 6 | 6 | 6
Participants
  All-causality TEAEs | 6 | 0 | 0 | 1 | 2 | 1 | 2 | 3 | 1 | 2
  Treatment-related TEAEs | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0

2. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities (Without Regard to Baseline [BL] Abnormality)
Description: Safety laboratory assessments included clinical chemistry, hematology, urinalysis, and other tests. Abnormality was determined at the investigator's discretion.
Time Frame: From BL to onsite Follow Up visit (up to 9 days after last dose of study intervention) (approximately up to 17 weeks)
Population: The analysis set included all participants randomly assigned to study intervention and who received a dose of study intervention. Participants with evaluable laboratory values were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | PF-07258669 0.1mg | PF-07258669 0.3mg | PF-07258669 1mg | PF-07258669 3mg | PF-07258669 10mg | PF-07258669 30mg | PF-07258669 100mg | PF-07258669 200mg | PF-07258669 300mg
Number analyzed (Participants) | 18 | 5 | 5 | 6 | 6 | 6 | 5 | 6 | 6 | 6
Participants | 14 | 5 | 3 | 4 | 4 | 6 | 5 | 6 | 6 | 3

3. Primary Outcome: Number of Participants With Change From BL in Vital Signs Data Meeting the Pre-defined Categorical Summarization Criteria
Description: Abnormality in change from BL in vital signs included: standing diastolic blood pressure (BP) increase and decrease from BL of >=20mmHg, standing systolic BP increase and decrease from BL of >=30mmHg, supine diastolic BP increase and decrease from BL of >=20mmHg, supine systolic BP increase and decrease from BL of >=30mmHg.
Time Frame: From BL to onsite Follow Up visit (up to 9 days after last dose of study intervention) (approximately up to 17 weeks)
Population: The analysis set included all participants randomly assigned to study intervention and who received a dose of study intervention. Participants with evaluable vital signs data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | PF-07258669 0.1mg | PF-07258669 0.3mg | PF-07258669 1mg | PF-07258669 3mg | PF-07258669 10mg | PF-07258669 30mg | PF-07258669 100mg | PF-07258669 200mg | PF-07258669 300mg
Number analyzed (Participants) | 18 | 5 | 5 | 6 | 6 | 6 | 5 | 6 | 6 | 6
Participants
  Standing diastolic BP increase >=20mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Standing diastolic BP decrease >=20mmHg | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Standing systolic BP increase >=30mmHg | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Standing systolic BP decrease >=30mmHg | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Supine diastolic BP increase >=20mmHg | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine diastolic BP decrease >=20mmHg | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Supine systolic BP increase >=30mmHg | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine systolic BP decrease >=30mmHg | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1

4. Primary Outcome: Number of Participants With Change From BL in Electrocardiogram (ECG) Data Meeting the Pre-defined Categorical Summarization Criteria
Description: ECG assessments inlcuded PR, QT, QTcF intervals and QRS complex. ECG abnormalities in change from BL included: PR interval BL >200msec and max >=25% increase from BL, or BL <=200msec and max >=50% increase from BL, QRS interval percent change from BL >=50%, QTcF change from BL >=30 and <=60msec, or change from BL >60msec.
Time Frame: From BL to onsite Follow Up visit (up to 9 days after last dose of study intervention) (approximately up to 17 weeks)
Population: The analysis set included all participants randomly assigned to study intervention and who received a dose of study intervention. Participants with evaluable ECG data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | PF-07258669 0.1mg | PF-07258669 0.3mg | PF-07258669 1mg | PF-07258669 3mg | PF-07258669 10mg | PF-07258669 30mg | PF-07258669 100mg | PF-07258669 200mg | PF-07258669 300mg
Number analyzed (Participants) | 18 | 5 | 5 | 6 | 6 | 6 | 5 | 6 | 6 | 6
Participants
  PR interval %change >=25/50% (BL >200msec and >=25% increase or BL <=200msec and >=50% increase) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS interval %change >=50% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF change >=30 and <=60msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF change >60msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically-significant Change From BL in Neurological Examination Findings
Description: The neurological exam consisted of assessment of higher cortical function, the cranial nerves, motor function, deep tendon reflexes, sensory exam, and coordination and gait, to the extent needed to assess the participant for any potential changes in neurological status, as determined by the investigator (or designee).
Time Frame: From BL to onsite Follow Up visit (up to 9 days after last dose of study intervention) (approximately up to 17 weeks)
Population: The analysis set included all participants randomly assigned to study intervention and who received a dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | PF-07258669 0.1mg | PF-07258669 0.3mg | PF-07258669 1mg | PF-07258669 3mg | PF-07258669 10mg | PF-07258669 30mg | PF-07258669 100mg | PF-07258669 200mg | PF-07258669 300mg
Number analyzed (Participants) | 18 | 5 | 5 | 6 | 6 | 6 | 5 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Maximum Observed Concentration (Cmax) of PF-07258669
Description: Cmax is the maximum observed plasma concentration.
Time Frame: At 0 (prior to dose), 0.17, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours post dose on Day 1 in Periods 1 to 4
Population: The PK parameter analysis population was defined as all participants randomly assigned to study intervention and who received a dose of study intervention, and had at least 1 of the PK parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-07258669 0.1mg | PF-07258669 0.3mg | PF-07258669 1mg | PF-07258669 3mg | PF-07258669 10mg | PF-07258669 30mg | PF-07258669 100mg | PF-07258669 200mg | PF-07258669 300mg
Number analyzed (Participants) | 5 | 5 | 6 | 6 | 6 | 5 | 6 | 6 | 6
nanogram per milliliter (ng/mL) | 0.8439 (13) | 3.053 (35) | 10.72 (40) | 26.48 (35) | 53.30 (24) | 188.1 (3) | 573.4 (45) | 1173 (41) | 1604 (64)

7. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of PF-07258669
Description: AUClast is the area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration.
Time Frame: At 0 (prior to dose), 0.17, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours post dose on Day 1 in Periods 1 to 4
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-07258669 0.1mg | PF-07258669 0.3mg | PF-07258669 1mg | PF-07258669 3mg | PF-07258669 10mg | PF-07258669 30mg | PF-07258669 100mg | PF-07258669 200mg | PF-07258669 300mg
Number analyzed (Participants) | 5 | 5 | 6 | 6 | 6 | 5 | 6 | 6 | 6
nanogram*hour per milliliter (ng*hr/mL) | 2.421 (13) | 7.826 (30) | 27.83 (27) | 75.84 (29) | 182.2 (16) | 584.8 (11) | 2148 (12) | 4013 (21) | 5764 (34)

8. Secondary Outcome: Area Under the Plasma Concentration Time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) of PF-07258669
Description: AUCinf is the area under the plasma concentration time profile from time 0 extrapolated to infinite time.
Time Frame: At 0 (prior to dose), 0.17, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours post dose on Day 1 in Periods 1 to 4
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-07258669 0.1mg | PF-07258669 0.3mg | PF-07258669 1mg | PF-07258669 3mg | PF-07258669 10mg | PF-07258669 30mg | PF-07258669 100mg | PF-07258669 200mg | PF-07258669 300mg
Number analyzed (Participants) | 5 | 5 | 6 | 6 | 6 | 5 | 6 | 6 | 6
nanogram*hour per milliliter (ng*hr/mL) | 2.659 (14) | 8.252 (28) | 28.55 (28) | 76.63 (28) | 183.0 (15) | 586.9 (11) | 2156 (12) | 4033 (21) | 6036 (32)

9. Secondary Outcome: Time for Cmax (Tmax) of PF-07258669
Description: Tmax is the time for Cmax.
Time Frame: At 0 (prior to dose), 0.17, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours post dose on Day 1 in Periods 1 to 4
Population: as for outcome 6
Measure: Median (Full Range); unit: hour
Arm/Group | PF-07258669 0.1mg | PF-07258669 0.3mg | PF-07258669 1mg | PF-07258669 3mg | PF-07258669 10mg | PF-07258669 30mg | PF-07258669 100mg | PF-07258669 200mg | PF-07258669 300mg
Number analyzed (Participants) | 5 | 5 | 6 | 6 | 6 | 5 | 6 | 6 | 6
hour | 1.00 [1.00 to 1.50] | 1.00 [0.500 to 1.00] | 0.750 [0.500 to 1.00] | 0.750 [0.500 to 1.00] | 1.00 [0.500 to 1.00] | 1.00 [1.00 to 1.00] | 1.00 [0.500 to 1.50] | 1.25 [1.00 to 2.00] | 1.00 [0.500 to 1.50]

10. Secondary Outcome: Terminal Half-life (t1/2) of PF-07258669
Description: t1/2 is the terminal half-life.
Time Frame: At 0 (prior to dose), 0.17, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, and 48 hours post dose on Day 1 in Periods 1 to 4
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF-07258669 0.1mg | PF-07258669 0.3mg | PF-07258669 1mg | PF-07258669 3mg | PF-07258669 10mg | PF-07258669 30mg | PF-07258669 100mg | PF-07258669 200mg | PF-07258669 300mg
Number analyzed (Participants) | 5 | 5 | 6 | 6 | 6 | 5 | 6 | 6 | 6
hour | 2.508 (0.92446) | 3.828 (0.92253) | 4.572 (0.93360) | 5.013 (0.52812) | 5.558 (0.78987) | 6.698 (1.6508) | 6.415 (1.5912) | 6.880 (1.9697) | 12.99 (10.045)

ADVERSE EVENTS:
Time Frame: From first dose of study intervention (Day 1) to telephone Follow Up (28-35 days after lase dose of study intervention) (approximately up to 20 weeks)
Description: SAEs and nonserious AEs were recorded on the Case Report Form. SAEs were also reported on the Clinical Trial SAE report form to Pfizer Safety within 24h of awareness. The same event may appear as both an AE and SAE. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs/AEs.
Arm/Group | Pooled Placebo | PF-07258669 0.1mg | PF-07258669 0.3mg | PF-07258669 1mg | PF-07258669 3mg | PF-07258669 10mg | PF-07258669 30mg | PF-07258669 100mg | PF-07258669 200mg | PF-07258669 300mg
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/5 | 0/5 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/5 | 0/5 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/18 | 0/5 | 0/5 | 1/6 | 2/6 | 1/6 | 2/5 | 3/6 | 1/6 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo (N=18) | PF-07258669 0.1mg (N=5) | PF-07258669 0.3mg (N=5) | PF-07258669 1mg (N=6) | PF-07258669 3mg (N=6) | PF-07258669 10mg (N=6) | PF-07258669 30mg (N=5) | PF-07258669 100mg (N=6) | PF-07258669 200mg (N=6) | PF-07258669 300mg (N=6)
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Noninfective gingivitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT04628793/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT04628793/SAP_001.pdf